CLINICAL TRIAL: NCT04020640
Title: Infant Feeding Practices in Transition: Breast Milk Intake, Complementary Feeding and Body Composition During Infancy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Wanabhorn Tongchom, Principle investigator, Mahidol University
Other Study IDs: MU-IRB 2012/114.0712
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Breast Feeding
Keywords: human milk intake; dose-to-mother deuterium oxide; exclusive breastfeeding; predominant breastfeeding; partial breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exclusive breastfeeding (EBF): provision of breast milk only, allowing only receiving oral rehydration salts (ORS), drops and syrups (vitamins, minerals, medicines) as necessary
  Interventions: Other: no intervention
- Predominant breastfeeding (PBF): providing breast milk plus other liquids (water and water-based drinks, fruit juice) and ORS, drops and syrups (vitamins, minerals, medicines)
  Interventions: Other: no intervention
- Partial breastfeeding (PartBF): provision of breast milk plus infant formula or cow milk or other solid/semi-solid complementary foods
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Measure human intake using stable isotope technique
  Other Names: Observational study

SUMMARY:
Research Aim: We assessed human milk intakes of Thai infants during the first 6 months comparing exclusive (EBF), predominant (PBF) and partial (PartBF) breastfeeding.

Methods: One-hundred and ten apparently healthy Thai lactating mother-infant pairs were followed from birth. Human milk intakes were determined at 6 weeks, 3 and 6 months, using the DTM method. Daily energy and protein intakes were assessed using 3-day non-consecutive 24-hour recalls. Socio-demographic characteristics were collected using a questionnaire. For comparisons among breastfeeding practices, one-way ANOVA with Tukey's post hoc test was used for normally distributed data, or Kruskal-Wallis Test with Mann-Whitney U Test for not normally distributed data.

DETAILED DESCRIPTION:
Human milk intakes were comparable between the EBF and PBF infants during the first 6 months, and provided the sole source of energy and protein; infant formula largely replaced breast milk among PartBF infants.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy women aged 20-35 year
* Had pre-pregnancy BMI in the normal range (18.5-25 kg/m2)
* Planned to breastfeed their baby for at least 6 months
* Being full term infants (gestational age 37-42 weeks) and singleton
* Had normal birth weight (2,500 - 4,000 g)
* Signed written informed consent to participate in the study

Exclusion Criteria:

* Infant: preterm; twin; low and high birth weight; congenital diseases
* Mother: chronic diseases needed to get medicine and treatment; underweight and obesity
* Mother and baby did not stay together throughout 12 months of infant age

Ages: 2 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The mother-infant pairs were recruited at the Ratchaburi hospital and Health promoting hospital, Health promotion center region 5, both situated in Ratchaburi province, central Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2015-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
Human milk intake of Thai breastfed infants during the first 6 months using the dose-to-mother deuterium dilution method | 6 months
  assessed human milk intakes of Thai infants during the first 6 months comparing exclusive (EBF), predominant (PBF) and partial (PartBF) breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: WANABHORN TONGCHOM, PhD, Principal Investigator — Institute of Nutrition

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogelezang S, Santos S, van der Beek EM, Abrahamse-Berkeveld M, Duijts L, van der Lugt A, Felix JF, Jaddoe VWV. Infant breastfeeding and childhood general, visceral, liver, and pericardial fat measures assessed by magnetic resonance imaging. Am J Clin Nutr. 2018 Oct 1;108(4):722-729. doi: 10.1093/ajcn/nqy137. PMID 30107466
- [Derived] Tongchom W, Pongcharoen T, Judprasong K, Udomkesmalee E, Kriengsinyos W, Winichagoon P. Human Milk Intake of Thai Breastfed Infants During the First 6 Months Using the Dose-to-Mother Deuterium Dilution Method. Food Nutr Bull. 2020 Sep;41(3):343-354. doi: 10.1177/0379572120943092. Epub 2020 Aug 17. PMID 32799695